CLINICAL TRIAL: NCT06885684
Title: Developing Cognitive Control and Metacognition to Reduce the Functional Impact of Restricted and Repetitive Behaviors in Autism
Brief Title: Cognitive Control and Metacognition Training
Acronym: CoMeT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FP01034542
Record Dates: First submitted 2025-03-11; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Autism; Autism Spectrum Disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: biostatistician; eeg analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Control Training + Metacognition Coaching (Experimental): Intervention will be delivered individually in person. Cognitive Control (CC) Computer Training consists of four games that require multiple aspects of CC (flexible thinking, inhibitory control) and working memory. Each game has approximately 20 levels of increasing difficulty. Parameters that contribute to the difficulty and passing criteria are fixed, but children progress from level to level at their own pace. Metacognition Coaching employs manualized strategies that: meaningfully engage children with the training tasks; simplify tasks to make them more manageable; support sustained effort; emphasize key CC skills needed for tasks; provide coping strategies to reduce frustration associated with challenging aspects of the games; and use guided conversations to aid children with mastering each game. To support the needs of children with ASD, key concepts are described using consistent language and visual supports throughout training sessions.
  Interventions: Behavioral: Cognitive Control Training + Metacognition Coaching
- Waitlist (No Intervention): The waitlist group will continue with any ongoing interventions (treatment as usual) and will not initially receive the training program. At the end of the study, the waitlist group will be offered training.

INTERVENTIONS:
Behavioral: Cognitive Control Training + Metacognition Coaching — Computer training is delivered in person by a coach. Training consists of four games; each requires multiple aspects of cognitive control. Training levels progress in difficulty by increasing the number of items or simultaneous dimensions, decreasing the available response time, requiring greater accuracy, or adjusting the proportion of distractors or their complexity. Parameters that influence the difficulty of each level and passing criteria are fixed, but children progress from level to level at their own pace. Training is accompanied by manualized metacognition coaching to provide strategies to meaningfully engage with the tasks, simplify the tasks, support sustained effort, emphasize key cognitive control skills needed, provide coping strategies to reduce frustration associated with challenging aspects of the games, and use guided conversations to highlight metacognition.
  Arms: Cognitive Control Training + Metacognition Coaching

SUMMARY:
95 autistic children (ages 8-11yrs) will be randomly assigned to a novel computer-based Cognitive Control Training combined with Metacognition Coaching or to a comparison group that receives the intervention after a delay. Before and after intervention, electroencephalography (EEG) will be used to examine engagement of the target neural responses.

DETAILED DESCRIPTION:
Effective interventions to reduce the functional impact of core features of autism spectrum disorder (ASD) in school-aged children are critically needed. This study will test whether in-person computer training delivered individually by a coach engages an electroencephalographic (EEG) biomarker of cognitive control (N2 event-related potential [ERP] amplitude). Developing more effective cognitive control, metacognition, and working memory is predicted to enhance neural responses to conflicting information (i.e., a neural marker of effective cognitive control). The study will randomly assign 95 autistic children (ages 8-11yrs) to a novel computer-based Cognitive Control Training combined with Metacognition Coaching or to a waitlist control group. Before and after intervention, EEG will be used to examine engagement of the target neural responses. We expect the group assigned to Cognitive Control Training + Metacognition Coaching to exhibit significantly larger changes in N2 ERP amplitude in incongruent relative to congruent trials than the waitlist group. Before and after intervention, we will collect neural responses and behavioral measures of cognitive control and working memory.

ELIGIBILITY:
Inclusion Criteria:

* Children should be 8 to 11 years of age
* Children should have an existing diagnosis of an autism spectrum disorder, which will be confirmed using research measures and criteria
* Children must have general cognitive ability in the average range or above (above 80 using the Wechsler Abbreviated Scale of Intelligence-2 Full Scale IQ)
* Caregivers and children must be fluent in English or Spanish

Exclusion Criteria:

* Children must not have a known genetic condition related to autism (e.g., Fragile X)
* Children must not have medical conditions/injuries, exposure to substances, or significant deprivation with implications for the central nervous system or that require regular psychoactive medications that alter EEG responses (anticonvulsants, barbiturates) *
* Children must not have seizures or a seizure disorder (other than history of febrile seizures)
* Children must not have significant sensory or motor impairment or major physical abnormalities that would limit the ability to participate in table top or EEG testing, or make responding during computer activities difficult
* Children must not have a failed screening for colorblindness

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Flanker N2 ERP mean amplitude (primary measure of target engagement) | Baseline (Pre Training/Waitlist Phase) and at 15-17 Weeks (Post Training/Waitlist Phase)
  The flanker portion of the Child Attention Network Task (ANT) measures neural response to CC monitoring and inhibition. It includes 12 practice and 108 test trials. Each trial begins with a 150ms beep paired with a 450ms fixation cross at the center of the screen. Then, a target and flankers are presented for 2000ms. Congruent trials (50%) include a central target animal flanked by two animals on each side with the same orientation and size as the target. Incongruent trials (50%) are identical except that the target and flankers face opposite directions.
  Children use two buttons to show the direction each target is facing (50% left, 50% right) and receive feedback.

SECONDARY OUTCOMES:
The Change Task - Stop Signal Reaction Time | Baseline (Pre Training/Waitlist Phase) and at 15-17 Weeks (Post Training/Waitlist Phase)
  It has four test blocks with Go (75%) and Change trials (25%). Change trials consist of a visual signal to stop the dominant task (i.e., left/right button press) and change response (i.e., space bar). Individual differences in reaction time (RT) are controlled using the mean correct RT from the previous block; stop signals occur equally at 50, 200, 350, and 500ms before each child's RT. Stop signal reaction time (SSRT) is computed via the mean method and estimates the latency to inhibit a dominant response.
Dimensional Change Card Sort t-score | Baseline (Pre Training/Waitlist Phase) and at 15-17 Weeks (Post Training/Waitlist Phase)
  The National Institute of Health (NIH) Toolbox Dimensional Change Card Sort (DCCS) measures cognitive control set-shifting. Four blocks (practice, pre-switch, post-switch, and mixed) are presented on a tablet. In a pre-switch block of 5 trials, children sort by one dimension (e.g., color). If 80% of trials are correct, they sort by a different dimension (e.g., shape) for 5 post-switch trials. If children pass the post-switch block, they switch back and forth between dimensions for 50 mixed trials (80% 'dominant') presented in a pseudorandom order (with 2-5 dominant trials preceding each non-dominant trial). The dominant dimension is always the sorting dimension used in the post-switch block. Scoring is based on the number of trials administered and integrates both accuracy and RT in a single score.
List Sorting Working Memory Test t-score | Baseline (Pre Training/Waitlist Phase) and at 15-17 Weeks (Post Training/Waitlist Phase)
  The NIH Toolbox List Sorting Working Memory Test requires children to sort pictures of animals and food. Stimuli appear for 2s while the name of the stimulus is read by a recorded voice. Children must remember each stimulus in a series, mentally reorder them from smallest to largest, and say the names in the new order. The '1-list' section presents only one type of stimulus. In the '2-list' section, children must first sort by category (animal or food) and then size. Scoring combines total items correct across the 1- and 2-list sections.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Faja, PhD, Principal Investigator — Boston Children's Hospital / Harvard Medical School

IPD SHARING:
Plan to Share IPD: Undecided